CLINICAL TRIAL: NCT06941311
Title: Integrating the Youth Nominated Support Team (YST) With CBT for Black Youth With Acute Suicide Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); MiSide (Unknown); Children's Hospital of Michigan (Other)
Responsible Party: Principal Investigator, Cynthia Ewell Foster, Clinical Associate Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00225071; 5R34MH131722-02 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Suicide Prevention
Keywords: Black youth; Acute suicide risk; Youth Nominated Support Team; Cognitive Behavioral therapy for Suicide Prevention; Community Mental Health; Suicide prevention
MeSH Terms: conditions — Suicide Prevention | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study will recruit 6 youth and 6 parents/guardians, as well as up to 24 support individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBT for Suicide Prevention and the Youth-Nominated Support Team (Experimental): Participation will be 3 months.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Suicide Prevention (CBT-SP); Behavioral: Youth-Nominated Support Team

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Suicide Prevention (CBT-SP) — Clinicians will provide this specialized evidence-based mental health care. The study focuses on the acute phase of CBT-SP, which is 12 sessions. CBT-SP's goals are to reduce suicide risk factors, enhance coping, and prevent future suicidal behavior. Identifying the emotional, cognitive, behavioral, or familial processes that precede a suicide crisis is a major focus, which yields an individualized treatment plan. Each session lasts one hour and can be completed either in person or via a secure telehealth platform. Most youths will attend sessions on a weekly basis and therapists typically like to be in contact with parents as well.
Behavioral: Youth-Nominated Support Team — Youth will nominate up to 4 trusted adults. Following parental approval, Support Persons will attend an orientation session with their assigned intervention specialist, learn about the youth's difficulties, treatment plan, and receive ideas for supporting the youth. Support Persons will be asked to have contact with the youth each week for up to three months to offer emotional support, encourage participation in treatment, and support the youth's healthy behaviors. Support Persons will have weekly check-ins with their intervention specialist every week for the 3 months of the study. During these calls, Support Persons have an opportunity to discuss any questions or concerns they may have about the youth and how best to support them.

SUMMARY:
The investigators are modifying and testing the preliminary effectiveness and implementation of the combination of two psychosocial interventions, Cognitive Behavioral Therapy for Suicide Prevention (CBT-SP) and the computer-assisted version of the Youth-Nominated Support Team (eYST). This registration will be for Aim 2 and a pilot randomized clinical trial for Aim 3 will be registered separately.

In this phase of the study, CBT-SP+eYST will be tested in an initial open trial (number of youth=6) to examine its feasibility and acceptability. Investigators will recruit Black adolescents that come to an urban emergency department (ED) for suicidal thoughts and/or behaviors to receive the intervention in an outpatient community mental health agency. The study focuses on the acute phase of CBT-SP, which is 12 sessions. Participants will nominate up to 4 caring adults in the participants lives to serve as support persons. These support persons will attend an education/orientation session to learn more about their role and how to support the youth.

Youth will be assessed at baseline, 6 weeks, and 14 weeks. Parents will be assessed at baseline and 14 weeks. Support persons will be assessed at baseline and 14 weeks. Fidelity assessments will be completed by clinicians after each CBT-SP session, after the YST psycho-ed session, and weekly to document contact with the support team.

ELIGIBILITY:
Inclusion criteria for youth:

* Patients of any gender between the ages of 12 and 17 years
* Patients that are able to provide at least one verifiable contact for emergency or tracking purposes
* Eligible for care at MiSide
* Present to the ED with suicide risk (per protocol)
* Self-identify as Black (obtain from face sheet collected in triage)
* Willing and able to complete enrollment procedures
* Willing and able to provide signed and dated informed assent

Exclusion criteria for youth:

* Unable to be consented in English
* Do not have a parent/legal guardian available to provide consent
* Are not able to provide informed assent or to participate in the assessment due to significant agitation, psychosis, cognitive impairment, learning disability, or medical trauma
* Actively engaged in specialty mental health treatment

Parent/Guardian Inclusion Criteria:

* Adults 18 years old and older
* The parent or legal guardian of a youth participating in Aim 2
* Understand written and spoken English
* Willing and able to complete enrollment procedures
* Willing and able to provide signed and dated informed consent

Parent/Guardian Exclusion Criteria:

- Do not understand written and spoken English

Support Person Inclusion Criteria:

* Adults 18 years and older
* Understand written and spoken English
* Approved to serve as a support person by the parent/legal guardian

Support Person Exclusion Criteria:

* Do not understand written and spoken English
* Not approved to serve as a support person by the parent/guardian

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability - percent of eligible youth consented | Baseline
  The intervention will be considered acceptable if at least 50% of eligible youth choose to enroll in the study.
Feasibility - Mean number of support people | 6 weeks
  The intervention will be considered feasible if the mean number of support people per youth is at least 3.
Acceptability - Mean number of support person contacts | 14 weeks
  The intervention will be considered acceptable if the mean number of support person contacts with youth is at least 7.
Feasibility - Number of CBT-SP sessions attended | 14 weeks
  Number of CBT-SP sessions attended by youth

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ewell Foster, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Children's Hospital of Michigan (CHM) Emergency Department, Detroit, Michigan
  - MiSide, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Upload to National Institute of Mental Health (NIMH) Data Archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is completed and available according to NIMH Data Archive policy.
Access Criteria: Researchers can request de-identified data from the study contacts listed in the study.
URL: https://nda.nih.gov/